CLINICAL TRIAL: NCT06700460
Title: A Randomized Evaluation of Clinical Outcomes Following Bilateral Implantation of EVO+ ICL Lenses or Bilateral Wavefront-Optimized LASIK (EVOlve)
Brief Title: Measuring Outcomes of LASIK and EVO-ICL in Matched Populations
Acronym: EVOlve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KJF-726
Record Dates: First submitted 2024-11-15; First posted 2024-11-22 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: LASIK; EVO ICL; Myopia; Clinical Outcomes
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Intervention Model Description: All LASIK procedures in this study are to be Wavefront Optimized treatments. To ensure standardization of treatments within the LASIK cohort, Wavefront-Guided and Topography-Guided treatments are prohibited. The EX500 laser, an excimer laser, employes a 1050 Hz multidimensional active tracker, online optical pachymetry, an onboard nitrogen generator and a 500 Hz laser pulse frequency that enables the treatment of each D of myopia in 1.4 seconds. The EX500 laser will perform the wavefront refraction according to the user manual and MOP instructions.
  Refer to current approved EVO+ ICL Directions for Use (DFU) for surgical instructions.6 Study surgeons will use 2% HPMC OVD for EVO+ ICL surgery as recommended in the DFU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laser-assisted in Situ Keratomileusis (Active Comparator): LASIK-Wavefront Optimized
  Interventions: Device: Implantable Collamer Lens placement
- Implantable Collamer Lens placement (Active Comparator): EVO ICL
  Interventions: Device: Laser-assisted in Situ Keratomileusis

INTERVENTIONS:
Device: Laser-assisted in Situ Keratomileusis — LASIK
  Arms: Implantable Collamer Lens placement
Device: Implantable Collamer Lens placement — EVO ICL
  Arms: Laser-assisted in Situ Keratomileusis

SUMMARY:
Evaluating outcomes after bilateral implantation of ICLs or bilateral LASIK as treatment options for the correction or reduction of myopia with or without astigmatism.

DETAILED DESCRIPTION:
A randomized evaluation of clinical outcomes following bilateral implantation of EVO+ Visian™ Implantable Collamer™ Lenses or bilateral Wavefront-optimized LASIK as treatment options for the correction or reduction of myopia with or without astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Preoperatively the Investigator will evaluate each study subject and refer to the directions for use for EVO+ ICL and Wavefront-Optimized LASIK to confirm the subject's suitability to proceed with bilateral EVO+ ICL Implantation or bilateral Wavefront-optimized LASIK in accordance with the Investigator's standard of care for each procedure. To ensure similar characteristics across study subjects, the Investigator will also adhere to the following criteria for each group:

  1. Subjects ages 21 to 45 years old.
  2. Stable refractive error for at least one year (≤ 0.50 D change in refraction) or stability as determined by the Investigator.
  3. Myopia or myopia with astigmatism with spherical equivalent ranging from -3.00 D to ≤ -8.00 D (in the spectacle plane) and cylinder in the range of 0.00 D to 4.00 D (in the spectacle plane).
  4. Corrected distance visual acuity (CDVA) of 20/20 or better in each eye.
  5. Difference between cycloplegic refraction spherical equivalent (CRSE) and manifest refraction spherical equivalent (MRSE) of ≤0.75 D.
  6. Subjects must be able and willing to return for scheduled follow-up examinations after surgery.
  7. Subjects must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.

Exclusion Criteria:

* 1. Pregnant or nursing women, or those who plan to become pregnant over the course of this clinical study or has another condition with associated fluctuation of hormones that could lead to refractive changes.

  2. Dry eye syndrome that is unable to be controlled with ocular lubricant(s) or medication(s) and which may confound study outcomes in the opinion of the Investigator.

  3. Serious acute, chronic, or systemic, non-ophthalmic disease or illness that would increase the operative risk, confound the outcome(s) of the study or which may preclude study completion (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, uncontrolled diabetes, etc.), in the opinion of the Investigator.

  4. Ocular condition (other than high myopia) that may predispose the subject to future complications, in the opinion of the Investigator. For example:
  * Pigment dispersion,
  * History or clinical signs of iritis/uveitis,
  * History of previous ocular surgery,
  * Monocular subjects,
  * History or evidence of active or inactive corneal disease (e.g., herpes simplex keratitis, herpes zoster keratitis, recurrent corneal erosion syndrome, corneal dystrophy, etc.),
  * Evidence of retinal vascular disease,
  * Keratoconus or keratoconus suspect,
  * Glaucoma or glaucoma suspect by exam findings,
  * Ocular surface disease other than controlled dry eye syndrome. 5. Subjects who do not qualify for both study arms:
  * Bilateral Wavefront Optimized LASIK
  * Bilateral EVO+ ICL implantation

    6. Subjects who, in the judgment of the Investigator, present any emotional, physiologic, or anatomical condition which may preclude participation in this study or provide an inappropriate landscape for the intended study treatment.

    7. Participation in another clinical trial involving ocular procedures within the last 6-months.

    8. Other conditions or assessment that causes the subject to not be an acceptable candidate for treatment or study participation as clinically assessed and documented by the Investigator.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 month
  Uncorrected distance visual acuity and Corrected distance visual acuity
Manifest refractive spherical equivalent | 1 month
  Manifest refraction spherical equivalent (MRSE) is a measurement used in eye care to determine the overall refractive error of the eye, taking into account both nearsightedness or farsightedness (spherical component) and astigmatism (cylindrical component).
  It's calculated by adding the sphere power and half of the cylinder power
Abberometry (Higher Order Abberations and Corneal Performance Index) | 1 month
  Aberrometry is a technique used to measure the optical aberrations of the eye, including both lower-order aberrations (LOAs) and higher-order aberrations (HOAs).
  LOAs are the standard refractive errors, such as nearsightedness, farsightedness, and astigmatism, which can be corrected with glasses or contact lenses. HOAs, on the other hand, are more complex aberrations that affect the quality of vision, even if the LOAs are corrected. HOAs are caused by irregularities in the shape of the cornea or lens.
  They can cause a variety of visual symptoms, including blurry vision, glare, halos, and difficulty seeing at night
Objective Scatter Index | 1 month
  The Objective Scatter Index (OSI) is a measurement used in ophthalmology to assess the quality of the eye's optical media, particularly the cornea and lens.
  It quantifies the amount of light scatter within the eye, which can affect visual clarity and contrast sensitivity.
Contrast Sensitivity | 1 month
  Contrast sensitivity is the ability to distinguish between objects with varying degrees of contrast, especially in situations of low light or when objects have subtle differences in shading.
Tear Film Stability | 1 month
  Tear film stability refers to the ability of the tear film, a thin layer of fluid that covers the surface of the eye, to remain intact and maintain a smooth, even surface. This is essential for clear vision and healthy ocular surface.
Ocular Adverse Events in treated eyes/safety | 1 month
  Ocular adverse events (OAEs) are side effects that can occur in the eye after receiving a treatment, such as medication, surgery, or radiation therapy.
  These events can range from mild and temporary to severe and permanent.
Subjective Questionnaires and Open-Ended Questions | 1 month
  Subjective questionnaires and open-ended questions are two common methods used in research to gather qualitative data. They allow researchers to delve deeper into participants' thoughts, feelings, and experiences, providing rich insights that quantitative methods may not capture.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Kugler Vision, Omaha, Nebraska
  - Cleveland Eye Clinic, Cleveland, Ohio
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Vance Thompson Vision Clinic, Sioux Falls, South Dakota
  - Slade & Baker Vision, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Per PI

REFERENCES:
- [Background] Ngo W, Situ P, Keir N, Korb D, Blackie C, Simpson T. Psychometric properties and validation of the Standard Patient Evaluation of Eye Dryness questionnaire. Cornea. 2013 Sep;32(9):1204-10. doi: 10.1097/ICO.0b013e318294b0c0. PMID 23846405
- [Background] Hays RD, Mangione CM, Ellwein L, Lindblad AS, Spritzer KL, McDonnell PJ. Psychometric properties of the National Eye Institute-Refractive Error Quality of Life instrument. Ophthalmology. 2003 Dec;110(12):2292-301. doi: 10.1016/j.ophtha.2002.07.001. PMID 14644710
- [Background] Sanders DR, Doney K, Poco M; ICL in Treatment of Myopia Study Group. United States Food and Drug Administration clinical trial of the Implantable Collamer Lens (ICL) for moderate to high myopia: three-year follow-up. Ophthalmology. 2004 Sep;111(9):1683-92. doi: 10.1016/j.ophtha.2004.03.026. PMID 15350323
- [Background] Directions for Use, EVO Visian® ICL (Implantable Collamer® Lens)." Accessed April 1, 2024. https://edfu.staar.com/edfu/.
- [Background] Moshirfar M, Durnford K, Megerdichian A, Thomson A, Martheswaran T, West W Jr, McCabe S, Ronquillo Y, Hoopes P. Refractive Outcomes After LASIK for the Treatment of Mixed Astigmatism with the Allegretto WaveLight EX500. Ophthalmol Ther. 2022 Apr;11(2):785-795. doi: 10.1007/s40123-022-00472-4. Epub 2022 Feb 15. PMID 35167040
- [Background] U.S. Food and Drug Administration. "PMA-P030008: WAVELIGHT EXCIMER LASER SYSTEM. "Accessed.fda.gov, https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpma/pma.cfm?id=P030008S006. Accessed 01Apr2024.
- [Background] Meidani A, Tzavara C. Comparison of efficacy, safety, and predictability of laser in situ keratomileusis using two laser suites. Clin Ophthalmol. 2016 Aug 24;10:1639-46. doi: 10.2147/OPTH.S110626. eCollection 2016. PMID 27601880
- [Background] Du H, Zhang B, Wang Z, Xiong L. Quality of vision after myopic refractive surgeries: SMILE, FS-LASIK, and ICL. BMC Ophthalmol. 2023 Jun 26;23(1):291. doi: 10.1186/s12886-023-03045-6. PMID 37365492